CLINICAL TRIAL: NCT03402906
Title: Family-Clinician Collaboration to Improve Neglect and Rehabilitation Outcome After Stroke
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient funding
Sponsor: Kessler Foundation (Other)
Responsible Party: Principal Investigator, Peii Chen, Senior Research Scientist, Kessler Foundation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E-991-17
Record Dates: First submitted 2018-01-02; First posted 2018-01-18 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2023-11

CONDITIONS: Stroke; Spatial Neglect
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Family-Clinician Collaboration (Experimental): Participants are dyads of a stroke survivor and their family member. Family members will work closely with the Clinician to understand the status and goals of the stroke survivor, and family members will integrate Family-Mediated Treatment Procedures into their time spent with the stroke survivor at home.
  Interventions: Behavioral: Family-Clinician Collaboration Program

INTERVENTIONS:
Behavioral: Family-Clinician Collaboration Program — Family-mediated treatment activities and collaboration between clinician and family members
  Other Names: FCC

SUMMARY:
Spatial neglect may occur in patients who have had a stroke. People with spatial neglect often pay much more attention to one side of the body while ignoring the other side, even though they have no difficulty seeing. The purpose of this study is to evaluate the impact on stroke recovery, including spatial neglect, of the Family-Clinician Collaboration program, where a family member of a stroke survivor actively interacts with clinical staff members providing inpatient rehabilitation services to the stroke survivor.

DETAILED DESCRIPTION:
Spatial neglect (SN) frequently occurs in patients who have had a stroke. The problems caused by SN result in patients failing to attend to the space contralateral to the side of the stroke. This failure to attend to half of the patient's field may result in problems with perception, memory, action planning and navigation. These deficits hurt both the patients and their caregivers, and make it difficult for them to resume daily activities as they were before the stroke. More than half of the patients who had SN at admission still had it when discharged from an inpatient rehabilitation facility.

This study examines a new behavioral treatment, where the clinician and the caregiver work together to provide better treatment. The family members will engage in frequent meetings with clinicians, set goals, learn about SN and coping strategies and have the patient to perform easy, safe treatment exercises. The study will compare this Family-Clinician Collaboration with the inpatient treatment control. This study will compare the groups in measures of spatial neglect and independence in the patients and measures of caretaker burden and mental health in family members. Participants will also report on their overall opinions of the new treatment condition.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral right brain stroke
* Functionally independent before stroke
* Presence of spatial neglect (moderate to severe, will be confirmed during the screening session)
* Ability to follow instructions and understand verbal or written English
* Currently living with a family member who will be enrolled into the study as well

Exclusion Criteria:

* History of progressive neurological disorder
* History of a significant psychiatric disorder
* Living outside of 50-mile radius of Kessler Foundation (West Orange, NJ)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-09-30 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Spatial neglect assessment battery | Before and immediately after intervention
  Searching visual targets, writing, reading, drawing, and other tasks that require exploration of the person's surroundings.
  The primary outcome measure is the change between before and immediately after intervention.
Family caregiver wellness | Before and immediately after intervention
  Self-reported questionnaires regarding emotional status, caregiving stress and burden.
  The primary outcome measure is the change between before and immediately after intervention.

SECONDARY OUTCOMES:
FCC feedback | Immediately after intervention
  Semi-structured interview on the experience of the study participation
Spatial neglect assessment battery | 4 weeks after intervention
  Searching visual targets, writing, reading, drawing, and other tasks that require exploration of the person's surroundings.
  The outcome measure is the change between immediately after intervention and 4-week follow-up.
Family caregiver wellness | 4 weeks after intervention
  Self-reported questionnaires regarding emotional status, caregiving stress and burden.
  The outcome measure is the change between immediately after intervention and 4-week follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Peii Chen, PhD, Principal Investigator — Kessler Foundation
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States

REFERENCES:
- [Derived] Longley V, Hazelton C, Heal C, Pollock A, Woodward-Nutt K, Mitchell C, Pobric G, Vail A, Bowen A. Non-pharmacological interventions for spatial neglect or inattention following stroke and other non-progressive brain injury. Cochrane Database Syst Rev. 2021 Jul 1;7(7):CD003586. doi: 10.1002/14651858.CD003586.pub4. PMID 34196963